CLINICAL TRIAL: NCT00760916
Title: FREEDOM DR: An International, Multi-Center, 12-Week, Double Blind, Randomized, Placebo-Controlled, Parallel Group Study Followed by a 12-Week Open-Label Extension Study to Assess the Efficacy, Safety, and Dose Response of UT-15C SR in Subjects With Pulmonary Hypertension
Brief Title: FREEDOM DR: Oral Treprostinil in Combination With an Endothelin Receptor Antagonist (ERA) and/or a Phosphodiesterase-5 (PDE-5) Inhibitor or as Monotherapy for the Treatment of Pulmonary Arterial Hypertension (PAH)
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Study stopped prior to subject enrollment.
Sponsor: United Therapeutics (Industry)
Responsible Party: Brett Goetz, Associate Manager, Clinical Operations, United Therapeutics
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TDE-PH-303
Record Dates: First submitted 2008-09-25; First posted 2008-09-26 (Estimated); Last update posted 2013-01-30 (Estimated); Status verified 2013-01

CONDITIONS: Pulmonary Hypertension
Keywords: Pulmonary Arterial Hypertension
MeSH Terms: conditions — Hypertension, Pulmonary; Pulmonary Arterial Hypertension | interventions — treprostinil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Placebo (Placebo Comparator): placebo
  Interventions: Drug: Placebo
- UT-15C 0.25 mg (Active Comparator): UT-15C 0.25 mg
  Interventions: Drug: UT-15C 0.25 mg
- UT-15C 1 mg (Active Comparator): UT-15C 1 mg
  Interventions: Drug: UT-15C 1 mg
- UT-15C 5 mg (Active Comparator): UT-15C 5 mg
  Interventions: Drug: UT-15C 5 mg

INTERVENTIONS:
Drug: UT-15C 1 mg — UT-15C 1 mg
  Arms: UT-15C 1 mg
Drug: UT-15C 0.25 mg — UT-15C 0.25 mg
  Arms: UT-15C 0.25 mg
Drug: UT-15C 5 mg — UT-15C 5 mg
  Arms: UT-15C 5 mg
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This study is an international, multi-center, randomized, double-blind, placebo-controlled study in subjects with PAH who are currently receiving approved therapy for their PAH (i.e., endothelin receptor antagonist and/or phosphodiesterase-5 inhibitor)or as a monotherapy treatment. Study visits will occur at 4 week intervals for 12 weeks with the key measure of efficacy being the 6-minute walk test. Study procedures include routine blood tests, medical history, physical exams, disease evaluation, and exercise tests. At the end of the first 12-weeks, the patient will be un-blinded. Patients will continue with another 12-Week open label portion with visits occuring at 4-week intervals.

Patients who complete all assessments for 24-weeks will also be eligible to enter a 36 month open-label, extension phase study (FREEDOM - EXT).

DETAILED DESCRIPTION:
This study is an international, multi-center, randomized, double-blind, placebo-controlled study in subjects with PAH who are currently receiving approved therapy for their PAH (i.e., endothelin receptor antagonist and/or phosphodiesterase-5 inhibitor)or as a monotherapy treatment. Study visits will occur at 4 week intervals for 12 weeks with the key measure of efficacy being the 6-minute walk test. Study procedures include routine blood tests, medical history, physical exams, disease evaluation, and exercise tests. At the end of the first 12-weeks, the patient will be un-blinded. Patients will continue with another 12-Week open label portion with visits occuring at 4-week intervals.

Patients who complete all assessments for 24-weeks will also be eligible to enter a 36 month open-label, extension phase study (FREEDOM - EXT).

ELIGIBILITY:
Inclusion Criteria:

* Between 18 and 70 years of age, inclusive
* Body weight at least 50 kilograms
* PAH that is either idiopathic/familial; associated with repaired congenital systemic-to-pulmonary shunts (repaired ≥ 5 years); associated with collagen vascular disease; associated with HIV.
* Currently receiving an approved endothelin receptor antagonist and/or an approved phosphodiesterase-5 inhibitor for at least 90 days and on a stable dose for at least the last 30 days or not currently receiving approved PAH therapy.
* Previous testing (e.g., right heart catheterization, echocardiography) consistent with the diagnosis of PAH.
* Reliable and cooperative with protocol requirements.

Exclusion Criteria:

* Nursing or pregnant.
* Received a prostacyclin within the past 30 days.
* PAH due to conditions other than noted in the above inclusion criteria.
* History of uncontrolled sleep apnea, renal insufficiency, anemia, left sided heart disease, uncontrolled systemic hypertension, or parenchymal lung disease.
* Use of an investigational drug within 30 days of Baseline

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-12; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Change in six-minute walk distance from Baseline to Week 12 | 12 weeks

SECONDARY OUTCOMES:
Borg Dyspnea Score | 12 weeks
Clinical Worsening Assessment | 12 weeks
Dyspnea Fatigue Index | 12 weeks
Symptoms of PAH | 12 weeks
World Health Organization (WHO) Functional Class | 12 weeks
Trough 6-Minute Walk Distance | 12 weeks
Trough Borg Dyspnea Score | 12 weeks
Pro-B-type natriuretic peptide (Pro-BNP) | 12 weeks
Optional hemodynamic parameters | 12 weeks
Adverse events | 12 weeks
Clinical Laboratory parameters | 12 weeks
Electrocardiogram findings | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Laliberte, PharmD, Study Director — United Therapeutics
Locations (31):
- United States (26):
  - University of Alabama Birmingham, Birmingham, Alabama
  - West Los Angeles VA Healthcare Center, Los Angeles, California
  - UC Davis Medical Center, Sacramento, California
  - Stanford University, Stanford, California
  - Pulmonary Hypertension Clinic, Aurora, Colorado
  - University of Iowa Health Care, Iowa City, Iowa
  - Kansas University Medical Center, Kansas City, Kansas
  - Maine Medical Center, Portland, Maine
  - Tufts Medical Center, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Minnesota, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Washington University Hospital, St Louis, Missouri
  - Weill Cornell Medical Center, New York, New York
  - Columbia Presbyterian Medical Center, New York, New York
  - Mary M Parkes Center for Asthma, Allergy and Pulmonary Care - University of Rochester, Rochester, New York
  - Duke University Medical Center, Durham, North Carolina
  - University Hospitals of Cleveland, Cleveland, Ohio
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University, Columbus, Ohio
  - Lagacy Clinic Northwest, Portland, Oregon
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - University of Texas Southwestern, Dallas, Texas
  - Intermountain Medical Center, Murray, Utah
  - Inova Fairfax Hospital, Falls Church, Virginia
- Australia (3):
  - St. Vincent's Hospital, Sydney, New South Wales
  - Prince Charles Hospital, Brisbane
  - The Alfred Hospital, Melbourne
- Mexico (2):
  - Instituto Nacional de Cardiologia, Mexico City, Mexico City
  - Unidad de Investigacion Clinica en Medicina (UDICEM), Monterrey